CLINICAL TRIAL: NCT06427486
Title: Investigating the Potential Efficacy, Feasibility, and Acceptability of Parent Telecoaching Intervention on Children With Autism and Their Parents in Palestine: A Mixed-Method Pilot Randomized Controlled Trial
Brief Title: Telecoaching Intervention for Children With Autism and Their Parents in Palestine
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Arab American University (Palestine) (Other)
Responsible Party: Principal Investigator, Mohammad Salahat, Instructor/ Head of Speech, Language, and Hearing Disorders Department, Arab American University (Palestine)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Parent Telecoaching and ASD
Record Dates: First submitted 2024-05-18; First posted 2024-05-24 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Autism Spectrum Disorder
Keywords: telecoaching; Telehealth; Early intervention; Quality of life; parent's self-competency; Activities of daily living; occupational performance coaching
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: This is a mixed-method pilot randomized waitlist-controlled trial with two parallel groups: the telecoaching intervention group and the waitlist control group, and semi-structured interviews with intervention participants. The utilization of a waitlist control group enables the comparison of the potential effects of the intervention group with those of a control group while ensuring that parents in the wait-listed control group can have access to telecoaching intervention after the completion of the study. After completing telecoaching sessions, participants from the intervention group will be invited to participate in semi-structured interviews to explore their perceptions about the intervention. The reason for using a mixed method is to achieve a comprehensive understanding of telecoaching intervention (its feasibility, acceptability, and potential efficacy) and to explain findings by connecting information obtained from both designs.
Masking Description: The trial author responsible for enrolling participants will not have access to the concealed random allocation sequence. However, due to the nature of the intervention, blinding the treatment assigned to participants will not be feasible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Parent Telecoaching Intervention (Experimental): The telecoaching intervention will consist of eight weekly sessions, lasting between 40 minutes to one hour each, conducted through Zoom. Before the sessions begin, an initial assessment meeting will take place with each parent. The sessions will follow the occupational performance coaching (OPC) processes, which aim to enhance parents' problem-solving skills and promote children's participation. These processes include the Connect, Structure, and Share stages, focusing on active listening, goal-setting, and information exchange between the provider and the parent. A Casenote template will be used to organize these sessions.
  Interventions: Other: Parents Telecoaching Intervention
- Access to a web-based (sanadmed). (No Intervention): The Waitlist Control Group Intervention will have access to a web-based Autism resources called "Sanad Al-Haya". This resource provides general information and videos on Autism and how to manage specific needs such as sensory issues, social interaction, and activities of daily living. The resources are developed by the trial author in Arabic language. All participants are required to register on the Sanad platform and create an account in their child's name. If they wish, the waitlist control group will have the option to take parent telecoaching sessions after the intervention group has completed all sessions.

INTERVENTIONS:
Other: Parents Telecoaching Intervention — - Synchronous (Zoom platform) and Asynchronous coaching sessions for parents of children with autism.
  Arms: Parent Telecoaching Intervention

SUMMARY:
In Palestine, children with autism spectrum disorder and their parents face difficulties in receiving needed early intervention and rehabilitation services due to a lack of specialized professionals and centers, as well as cultural, political, geographical, and financial barriers. Parents also face difficulties in raising their children with autism in their homes as they lack knowledge about the disorder and the best interventions that can be used to help these children.

Parent telecoaching intervention, or what is called (distance coaching via technology) can help parents and their children with autism. However, no research exists studying the possibility of using this intervention with parents and their children in Palestine and if it can have positive results on both parents and children.

The goal of this trial is to learn if parent telecoaching intervention is feasible and acceptable to parents of children with autism in Palestine. It will also learn if this intervention has the potential to improve children's skills and increase parent's self-competency and quality of life. The main questions it aims to answer are:

* To what extent and in what ways is providing telecoaching intervention for parents of children with Autism in Palestine possible?
* How do parents see telecoaching intervention in terms of suitability, benefits, facilitators, and barriers?
* Does telecoaching intervention for parents have the potential to increase children's participation in daily activities that parents consider important?
* Does telecoaching intervention have the potential to enhance parents' self-competence and family quality of life? Researchers will compare parent telecoaching intervention to a web-based resource designed to provide parents with general information about autism to see if parent telecoaching intervention works to help children with autism and their parents more than the free autism resources provided on the website.

Participants will:

* Take a telecoaching intervention (eight sessions over eight weeks, each session lasts one hour) or use the information provided on the website about autism.
* Apply the planned strategies with their children during the week and record their work using videos or by filling out a form to be reviewed at the beginning of each session.

DETAILED DESCRIPTION:
A purposive sampling technique will be used to recruit children with Autism Spectrum Disorder and their parents/caregivers who live in the West Bank districts. Two recruitment strategies will be used to invite participants from various districts in the West Bank. The first will involve approaching a third party, the Superhero Autism Foundation, to distribute invitation packages to potential eligible participants based on the provided inclusion and exclusion criteria. This foundation has been chosen as it has access to a vast dataset of children with autism across the West Bank. The second strategy will involve advertising flyers on social media and patient organization websites. Those who wish to participate will be asked to send their signed reply slip form to the trial's author using the contact information provided (email or WhatsApp). After that, they will be contacted by phone to screen their eligibility. Parents who meet the eligibility criteria will be informed that an initial meeting with each one of them will be conducted to explain the purpose of the trial further, check their willingness to be randomized, answer any questions they may have, confirm their consent to participate, agree on the first assessment meeting date and time which will be done before randomization, and discuss the schedule of the subsequent telecoaching sessions.

Sample size: A pilot randomized trial typically does not require a sample power calculation. However, as a rule of thumb, at least 30 participants will be needed for a pilot Randomized Controlled Trial. To address a potential attrition rate of 10%, 40 parent-child dyads (20 in each group) will be recruited.

Randomisation: The study will employ a stratified block randomization method to assign parents to either the telecoaching intervention group or the waitlist control group in a 1:1 ratio. Once baseline assessments are completed with eligible participants who have consented to participate, a screening number will be allocated to each parent, and the child's autism symptoms score will be recorded. This score will be categorized as <60 or ≥60 using the Autism Treatment Evaluation Checklist. The assigned screening number and the child's autism severity score for each participant will then be sent to a non-study member, a lecturer in the Occupational Therapy Department, who will conduct the allocation and randomization process based on predetermined block sizes of four using a computer-generated random sequence. Stratification will be conducted based on autism severity categorized as <60 or ≥60. This method is chosen to ensure an equal distribution of participants in each group and to minimize the impact of children's autism severity. The trial author responsible for enrolling participants will not have access to the concealed random allocation sequence. However, due to the nature of the intervention, blinding the treatment assigned to participants will not be feasible. All data from randomized participants will be recorded in a Case Report Form (CRF). Participants will be informed of the randomization outcome via phone contact.

Quantitative Data Analysis:

The Statistical Package for the Social Sciences (SPSS) version 26 will be used to conduct all statistical analyses.

Descriptive statistics will be used to analyze the following:

* Feasibility Criterions (1,3, 4, 6): eligibility, retention, provider intervention fidelity, and adverse event (if it occurs).
* Participants' demographic data will be analysed using percentages, mean, and standard deviation).
* The commonalities among family-specified goals on the Canadian Occupational Performance Measure (COPM).

Inferential statistics (Potential efficacy of Parent telecoaching intervention):

A t-test will be used to examine changes in means from pre-to-post-tests (between and within groups).

Qualitative Analysis (Acceptability, benefits, facilitators and barriers):

The recorded interviews will be analyzed using six iterative steps: (1) familiarization, (2) initial coding, (3) theme identification, (4) theme review, (5) theme definition and naming, and (6) report production. The trial author and a colleague will review and create initial codes, revisit the full transcriptions, and search for themes using the codes. They will meet multiple times to ensure theme names accurately describe the reports.

ELIGIBILITY:
Inclusion Criteria:

* Parents are the primary caregivers spending most of the intervention period with their child
* Parents are at least 18 years old and able to provide informed consent
* Parents have access to mobile devices such as phones, tablets or computers with Zoom software and a stable internet connection
* The children are between the ages of 3 and 6 years old and have a confirmed ASD diagnosis from a psychiatrist or pediatrician.
* Children with ASD and other comorbid conditions are also eligible to participate.

Exclusion Criteria:

* Adolescents and older adults with ASD.

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-03-02 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Canadian Occupational Performance Measure | Baseline, pre-intervention
  is used to help parents identify and prioritize the goals they want their child to achieve in the domains of self-care, productivity, and leisure. The tool involves parents rating each identified goal on a scale of 1 to 10, with 1 indicating that the goal is not important and 10 indicating that it is extremely important. From the list of identified goals, parents select the top five that they want to work on during the intervention. Parents then rate their child's performance and their satisfaction with that performance on a scale of 1 to 10, with 1 indicating that they are not satisfied and 10 indicating that they are extremely satisfied. This helps to measure changes in parents' perception of their child's performance and their satisfaction with that change from pre-test to post-test. The COPM has demonstrated sound psychometric properties with parents of children with disabilities, including construct validity and criterion validity.

SECONDARY OUTCOMES:
The 36-Item Short Form Health Survey questionnaire (SF-36) | Baseline, pre-intervention
  is used to evaluate the quality of life of parents using a 36-item Likert-type scale that measures eight domains (general health, physical role limitation, role limitation arising from emotional issues, physical functioning, vitality, mental health, bodily pain, and social function). The SF-36 questionnaire provides scores ranging from 0 to 100, with higher scores indicating better QoL. The questionnaire has been translated into Arabic, culturally validated, and utilized in research aimed at investigating the QoL of parents of children who have autism.
Parental Competence Scale for Children with Autism Spectrum Disorder | Baseline, pre-intervention
  This is a 29-item Arabic scale that measures parental competence for children with ASD. Each item has a 5-point rating scale. The scale is used to rate statements based on whether parents agree or disagree with them. A score of 5 is given to "Strongly Agree," while a score of 1 is given to "Strongly Disagree" for positive statements. For negative statements, the score is reversed. The minimum score is 29, while the maximum is 145. The validity of the tool was ensured by specialized staff in education psychology, and the reliability of the tool was tested demonstrating acceptable value (Cronbach Alpha 0.89).
Autism Treatment Evaluation Checklist (ATEC) | Baseline, pre-intervention
  This tool is used to identify the severity of autism and assess the effectiveness of interventions and treatments. It comprises of 77 questions that are divided into four categories: speech/language/communication (14 questions), sociability (20 questions), sensory/cognitive awareness (18 questions), and health/physical/behavior (25 questions). Parents or caregivers are responsible for completing the checklist, and lower scores indicate milder symptoms. The ATEC has been translated into Arabic and validated, revealing good internal consistency (a= 0.84), content validity (90% among referees), and construct validity

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Salahat, PhD, Principal Investigator — Arab American University (Palestine)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aschbrenner KA, Kruse G, Gallo JJ, Plano Clark VL. Applying mixed methods to pilot feasibility studies to inform intervention trials. Pilot Feasibility Stud. 2022 Sep 26;8(1):217. doi: 10.1186/s40814-022-01178-x. PMID 36163045
- [Background] Dahl-Popolizio S, Carpenter H, Coronado M, Popolizio NJ, Swanson C. Telehealth for the Provision of Occupational Therapy: Reflections on Experiences During the COVID-19 Pandemic. Int J Telerehabil. 2020 Dec 8;12(2):77-92. doi: 10.5195/ijt.2020.6328. PMID 33520097
- [Background] Dunn W, Little LM, Pope E, Wallisch A. Establishing Fidelity of Occupational Performance Coaching. OTJR (Thorofare N J). 2018 Apr;38(2):96-104. doi: 10.1177/1539449217724755. Epub 2017 Aug 18. PMID 28821218
- [Background] Efird J. Blocked randomization with randomly selected block sizes. Int J Environ Res Public Health. 2011 Jan;8(1):15-20. doi: 10.3390/ijerph8010015. Epub 2010 Dec 23. PMID 21318011
- [Background] Eldridge SM, Chan CL, Campbell MJ, Bond CM, Hopewell S, Thabane L, Lancaster GA; PAFS consensus group. CONSORT 2010 statement: extension to randomised pilot and feasibility trials. Pilot Feasibility Stud. 2016 Oct 21;2:64. doi: 10.1186/s40814-016-0105-8. eCollection 2016. PMID 27965879
- [Background] Little LM, Pope E, Wallisch A, Dunn W. Occupation-Based Coaching by Means of Telehealth for Families of Young Children With Autism Spectrum Disorder. Am J Occup Ther. 2018 Mar/Apr;72(2):7202205020p1-7202205020p7. doi: 10.5014/ajot.2018.024786. PMID 29426380
- [Background] Whitehead AL, Julious SA, Cooper CL, Campbell MJ. Estimating the sample size for a pilot randomised trial to minimise the overall trial sample size for the external pilot and main trial for a continuous outcome variable. Stat Methods Med Res. 2016 Jun;25(3):1057-73. doi: 10.1177/0962280215588241. Epub 2015 Jun 19. PMID 26092476
- [Background] Yazdani S, Capuano A, Ghaziuddin M, Colombi C. Exclusion Criteria Used in Early Behavioral Intervention Studies for Young Children with Autism Spectrum Disorder. Brain Sci. 2020 Feb 13;10(2):99. doi: 10.3390/brainsci10020099. PMID 32069875